CLINICAL TRIAL: NCT02590055
Title: Phase 2 Study of Gemcitabine and Docetaxel Combination Chemotherapy in Patients With Carcinoma of Unknown Primary
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Su Jin Lee, MD, PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-03-083
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Carcinoma of Unknown Primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention arm (Experimental): D1, 8 Gemcitabine 1000mg/m2 IV over 30 minutes D1, 8 Docetaxel 35mg/m2 IV over 1hr
  Interventions: Drug: gemcitabine/docetaxel combination

INTERVENTIONS:
Drug: gemcitabine/docetaxel combination

SUMMARY:
It's a phase 2, single arm study of gemcitabine an docetaxel combination in patients with carcinoma of unknown primary.

ELIGIBILITY:
Inclusion Criteria:

* 1. age>=20 2. pathologically confirmed patients with carcinoma of unknown primary 3. unfavorable type of CUP 4. ECOG PS 0-2 5. more than 1 evaluable lesion 6. life expectancy > 12 weeks 7. no prior history of chemotherapy 8. more than 2 weeks after surgery or radiotherapy 9. proper organ function 10. written informed consent

Exclusion Criteria:

* 1. favorable group CUP

  * squamous cell carcinoma in the cervical or inguinal LN only women with axillary LN metastasis only women with peritoneal carcinomatosis only well-differentiated neuroendocrine tumors poorly-differentiated tumors with midline tumor or elevated human HCG/AFP men with adenocarcinoma and elevated PSA 2. severe, unstable heart disease 3. uncontrolled systemic disease (DM, HTN, hypothyroidism, infection...) 4. pregnant or feeding women 5. current CNS tumor (except total removal or WBRT/GKS done)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | one year after later patients enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Su Jin Lee, MD, PhD, Principal Investigator — department of medicine, Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea